CLINICAL TRIAL: NCT04810104
Title: Parkinson's Disease With Mild Cognitive Impairment Treated With Nicotinic Agonist Drug
Acronym: PD-MIND
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Delays due to COVID
Sponsor: King's College London (Other)
Collaborators: Helse Stavanger HF (Other Government); Michael J. Fox Foundation for Parkinson's Research (Other); Parkinson's UK (Other); AstraZeneca (Industry); Masaryk University (Other); Norges Parkinsonforbund, Norway (Unknown); University of Exeter (Other); Stichting Lygature (Unknown); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD-MIND; 2019-002423-15 (EudraCT Number)
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
Keywords: Parkinson's Disease; Mild Cognitive Impairment; Cognition
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — spiro(1-azabicyclo(2.2.2)octane-3,2'(3H)-furo(2,3-b)pyridine)

STUDY DESIGN:
Intervention Model Description: This is a randomised, double-blind, placebo-controlled, parallel-group, phase 2a study of AZD0328, a selective α7 nicotinic receptor agonist, in PD-MCI.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active drug: AZD0328 (Experimental): Participants will receive AZD0328 capsules for oral administration.AZD0328 is a selective α7 nicotinic receptor agonist, The total daily dosage of AZD0328 is 1mg per day; administered as 0.5mg twice daily / BID. The study treatment period is 12-weeks.
  Interventions: Drug: AZD0328
- Placebo (Placebo Comparator): Participants will receive identical-appearing placebo capsules for oral administration.Participants will be instructed to take 2 capsules in the morning and 2 capsules in the evening for a 12-week period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0328 — Active study drug
  Arms: Active drug: AZD0328
Drug: Placebo — Non-active study drug
  Arms: Placebo

SUMMARY:
To test for the first time the potential of a nicotinic agonist on cognitive symptoms in people with mild cognitive impairment (MCI) in Parkinson's disease (PD), referred to as PD-MCI.

DETAILED DESCRIPTION:
There is an unmet clinical need to treat PD-MCI. As outlined previously, PD-MCI is common, has important clinical consequences, and there is currently no available treatment. Moreover, the underlying pathology of cognitive impairment in PD indicates that nicotinic agonists may be particularly relevant for this condition. This is a randomised, double-blind, placebo-controlled, parallel-group, phase 2a study of AZD0328, a selective α7 nicotinic receptor agonist, in PD-MCI. The study is an international, multi-centre study, which will take place across sites in Europe.

PD-MIND will for the first time test the potential of a nicotinic agonist on cognition in PD-MCI. The primary outcome is attention, as it is a key cognitive domain in the PD-MCI profile and most likely to be affected by a α7 nicotinic agonist. Exploratory outcome measures will guide decisions on the design and conduct of future larger Phase 3 trials. Qualifying participants will be randomly assigned at baseline to either receive 0.5mg twice a day (bis in die, BID) of AZD0328 or placebo for 12 weeks. A total of 160 participants with PD-MCI will be enrolled to the study: 80 in the active (AZD0328) group and 80 in the control (placebo) group. Participants will undertake face-to-face assessments at screening, baseline, and then 3- 6- and 12- weeks after beginning study treatment (see Figure 2 for trial design overview). A subset of 90 participants will also undergo an MRI biomarker component prior to study drug administration and at study end.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 to 80 years (inclusive) at time of consent
* Duration of motor symptoms of at least 1 year
* Hoehn and Yahr stage between 1 and 3 (inclusive) in ON state
* Diagnosis of PD according to United Kingdom (UK) Brain Bank criteria
* Score on Clinical Dementia Rating (CDR) scale = 0.5
* Diagnosis of PD-MCI according to MDS PD-MCI, Level I criteria
* Duration of cognitive impairment of at least 3 months (to distinguish from mild delirium)

Exclusion Criteria:

* Insufficient fluency in English or local language to complete assessments
* Severe visual or auditory impairment that may interfere with participant's ability to complete assessments
* Unable to provide informed consent at screening visit
* Participation in a clinical study involving an investigational drug within 4 months prior to screening
* Smoking (cigarettes, pipes, cigars, e-cigarettes etc.) or use of smokeless tobacco products (chewing / dipping tobacco, snuff etc.) or anti-smoking nicotine containing products (patches/gum/sprays etc.), within the last 12 weeks
* HADS depression subscale score ≥ 11
* History of deep brain stimulation or other neurosurgical procedure
* Diagnosis of dementia, including Parkinson's disease dementia (PDD) or Dementia with Lewy Bodies (DLB).
* Diagnosis of schizophrenia, bipolar disorder or other psychotic disorder
* Malignant neoplasms within 3 years of screening (except for basal or squamous cell carcinoma of the skin); or had curative surgery/treatment and has been free of malignancy for at least 12 months)
* Any medical condition that in the opinion of the investigator may be contributing to cognitive impairment, above and beyond that caused by the participant's PD,
* Current evidence of any other medical condition not stably or adequately controlled, and which in the opinion of the investigator may affect participant safety or study participation
* Using any prohibited medications or permitted medications that do not meet stable dosing regimen requirements, as specified in section 5.7
* Clinically significant vital sign or ECG measure at screening or baseline visit, that in the opinion of the investigator would prevent participant from safely participating in this study
* Clinically significant clinical laboratory result from screening visit, that in the opinion of the investigator would prevent participant from safely participating in this study
* Significant renal function impairment as indicated by estimated glomerular filtration rate (eGFR) < 45ml/min); Note: The eGFR is calculated using a formula derived from the Modification of Diet in Renal Disease Study (MDRD formula): eGFR= [186.3 x (Creatinine/88.4)-1.154 x (Age)-0.203] x [0.742 if female] x [1.210 if black]
* Unable to complete computerised cognitive test battery
* Marked cerebrovascular disease from MRI or CT scan within last 12 months (defined as Fazekas scale ≥ grade 3)
* Females who are breast-feeding
* Female participants assessed as being of child-bearing potential that have a positive pregnancy test at screening or baseline
* The participant does not understand or agree to comply with the contraception or reproductive requirements of the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in Attentional Intensity Index composite factor score from baseline to week 12 | From baseline to week 12 (end of treatment period).
  The Attentional Intensity Index composite factor score combines the speed scores from the three attention tasks (simple reaction time, choice reaction time and digit vigilance), and has been validated using factor analysis. The measure reflects the ability to focus attention and process information.

SECONDARY OUTCOMES:
Change in Attentional Intensity Index composite factor score from baseline to week 6 | From baseline to week 6 (mid-point of treatment period)
  The Attentional Intensity Index composite factor score combines the speed scores from the three attention tasks (simple reaction time, choice reaction time and digit vigilance), and has been validated using factor analysis. The measure reflects the ability to focus attention and process information.
Change in Sustained Attention Index composite factor score from baseline to week 6 and week 12 | From baseline to week 6 (mid-point of treatment period) and week 12 (end of treatment period)
  The Sustained Attention Index composite factor score combines the accuracy scores from choice reaction time and digit vigilance tasks, and reflects the ability to sustain attention and ignore distraction.
Change in Working Memory Index composite factor score from baseline to week 6 and week 12 | From baseline to week 6 (mid-point of treatment period) and week 12 (end of treatment period)
  The Working Memory Index composite factor score combines the accuracy scores from the two working memory tasks to form this measure, which reflects the capability of holding information in working memory.
Change in Episodic Memory Index composite factor score from baseline to week 6 and week 12 | From baseline to week 6 (mid-point of treatment period) and week 12 (end of treatment period)
  The Episodic Memory Index composite factor score combines the verbal recall and recognition tasks with visual recognition. It reflects the longer term memory capability, like how well someone can remember a short story or what they had for dinner last night, or what they did on their last birthday.
Change in Memory Speed Retrieval Index composite factor score from baseline to week 6 and week 12 | Fom baseline to week 6 (mid-point of treatment period) and week 12 (end of treatment period)
  The Memory Speed Retrieval Index composite factor score combines the speed scores from the two working memory tasks and the picture recognition task. Factor analysis has established that the speed of retrieval from working memory and episodic memory load on a common factor, and the score reflects the time taken to successfully retrieve information held in memory.
Change in MoCA score from screening to week 12 | From screening to week 12 (end of treatment period)
  The Montreal Cognitive Assessment (MoCA) assesses 8 cognitive areas: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation. Scores range from 0 to 30, with lower scores indicative of greater cognitive impairment.
Change in Sustained Attention Index composite factor score from week 12 to week 16 | From week 12 (end of treatment period) to week 16 (4 weeks after end of study medication dosing)
  The Sustained Attention Index composite factor score combines the accuracy scores from choice reaction time and digit vigilance tasks, and reflects the ability to sustain attention and ignore distraction.
Change in Working Memory Index composite factor score from week 12 to week 16 | From week 12 (end of treatment period) to week 16 (4 weeks after end of study medication dosing)
  The Working Memory Index composite factor score combines the accuracy scores from the two working memory tasks to form this measure, which reflects the capability of holding information in working memory.
Change in Episodic Memory Index composite factor score from week 12 to week 16 | From week 12 (end of treatment period) to week 16 (4 weeks after end of study medication dosing)
  The Episodic Memory Index composite factor score combines the verbal recall and recognition tasks with visual recognition. It reflects the longer term memory capability, like how well someone can remember a short story or what they had for dinner last night, or what they did on their last birthday.
Change in Memory Speed Retrieval Index composite factor score from week 12 to week 16 | From week 12 (end of treatment period) to week 16 (4 weeks after end of study medication dosing)
  The Memory Speed Retrieval Index composite factor score combines the speed scores from the two working memory tasks and the picture recognition task. Factor analysis has established that the speed of retrieval from working memory and episodic memory load on a common factor, and the score reflects the time taken to successfully retrieve information held in memory.
Change in MDS-UPDRS Part III motor examination subscale score from baseline to week 12 | From baseline to week 12 (end of treatment period)
  Part III of the Movement Disorder Society's (MDS) Unified Parkinson's Disease Rating Scale (UPDRS), is a motor examination and objective assessment of parkinsonism. This is based on 18 items assessed by the investigator, resulting in 33 scores by location and lateralization. These 33 scores are ratings on severity: from 0 (normal) to 4 (severe).The MDS-UPDRS-III total score ranges from 0 to 132, with higher scores indicative of more severe motor and functional impairment.
Change in total score from the Non-Motor Symptom Scale from baseline to week 12 | From baseline to week 12 (end of treatment period)
  The Non-Motor Symptoms Scale (NMSS) is a 30-item rater-based scale to assess a wide array of non-motor symptoms in patients with Parkinson's disease. The NMSS measures severity (scored 0 - 3) and frequency (scored 1 - 4) of non-motor symptoms across nine dimensions. The NMSS total score ranges from 0 to 360, with higher score indicative of worse non-motor symptoms.
Change in total score from the 39-item Parkinson's Disease Questionnaire from baseline to week 12 | From baseline to week 12 (end of treatment period)
  The 39-item Parkinson's Disease Questionnaire (PDQ-39) is a health-related quality-of-life questionnaire. The questionnaire contains 39 self-reported items on eight domains: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and body discomfort. Each item is scored on 5-point Likert-type scale from 0 (never) - 4 (always), over the past month. The PDQ-39 total score is 156: the lower the score reflects a better health-related quality-of-life.
Change in MCI-CGIC from baseline to week 12 | From baseline to week 12 (end of treatment period)
  The MCI-adjusted Clinical Global Impression of Change (CGIC) score is generated in the context of a semi-structured interview and is an indication of the change in the participant's global status, cognition, behaviour, and functional abilities on a 7-point scale, with the best score being 'marked improvement' and the worst being 'marked worsening.'
Change in depression and anxiety subscale scores from the HADS from baseline to week 12 | From baseline to week 12 (end of treatment period)
  The Hospital Anxiety and Depression Scale (HADS), has an anxiety (score 0 - 21) and a depression subscale (0 - 21), with higher subscales scores indicative of greater levels of depression / anxiety
Incidence, nature and severity of AEs and SAEs during treatment period | From baseline to week 12 (end of study treatment)
  Adverse Events (AEs) and Serious Adverse Events (SAEs)
Incidence of dosage reduction or treatment discontinuation during treatment period | From baseline to week 12 (end of study treatment)
  Dosage reduction or treatment discontinuation
Incidence of clinically significant changes or abnormal electrocardiogram (ECG) assessments, vital sign measurements and clinical laboratory values during treatment period | From baseline to week 12 (end of study treatment)
  Clinically significant laboratory values or vital sign measurements
Changes in whole-brain and regionally specific brain volumes from baseline/screening to week 12 | From screening/baseline (pre-medication dosing) to week 12 (end of study treatment)
  MRI scans
Changes in whole-brain perfusion as well as perfusion in regions of interests (ROIs) from baseline/screening to week 12 | From screening/baseline (pre-medication dosing) to week 12 (end of study treatment)
  MRI scans
Changes in functional resting-state connectivity of the large-scale cognitive brain networks from baseline/screening to week 12 | From screening/baseline (pre-medication dosing) to week 12 (end of study treatment)
  MRI scans

OTHER OUTCOMES:
Screening/Baseline whole-brain and regionally specific brain volumes as predictors of treatment response | At screening/baseline (pre-medication dosing)
  MRI scans
Screening/Baseline whole-brain perfusion as well as perfusion in ROIs as predictors of treatment response | At screening/baseline (pre-medication dosing)
  MRI scans
Screening/Baseline functional resting-state connectivity of the large-scale cognitive brain networks as predictors of treatment response | At screening/baseline (pre-medication dosing)
  MRI scans
Placebo-controlled change in levels of exploratory blood-based biomarkers for neuroprotection and/or disease modification changes | At baseline and week 12
  Blood-based biomarkers (e.g. cytokines, amyloid species, tau and alpha-synuclein)
Change in levels of study medication in blood from baseline to week 12 | From baseline to week 12 (end of treatment period)
  Levels of study medication in blood

CONTACTS AND LOCATIONS:
Overall Officials: Dag Aarsland, PhD, Study Director — King's College London; Stavager Univeristy Hospital

IPD SHARING:
Plan to Share IPD: No